CLINICAL TRIAL: NCT05820438
Title: Evaluation of Masticatory Muscle Activity in Pediatric Patients Undergoing Rapid Maxillary Expansion: a Prospective Study.
Brief Title: Evaluation of Masticatory Muscle Activity in Pediatric Patients Undergoing Rapid Maxillary Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-EMGRME
Record Dates: First submitted 2023-03-14; First posted 2023-04-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Maxillar Hypoplasia
MeSH Terms: conditions — Retrognathia | interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients requiring orthopedic treatment with Rapid Maxillary Expander (Experimental): Patients will be treated with Rapid Maxillary Expander with two bands on the upper first permanent molars or upper second primary molars (depending on the eruptive stage of the patient). The screw will be activated according to clinitian's indication until a transverse overcorrection of 2 mm is achieved in the first permanent molars. When the active disjunction phase is completed, the screw will be blocked out with a metal legature and the patient will wear the cemented RME for retentions at least for six months.
  Interventions: Device: Electromyography

INTERVENTIONS:
Device: Electromyography — Disposable bipolar surface electrodes will be used.
  The patient's skin will be clean with cotton gauze soaked in alcohol before electrodes placement to reduce skin impedance. The operator will palpate the muscle belly while the patient clenches his teeth and will position surface electrodes in parallel to the muscular fibres.Doing so the position of the electrodes results as follows:
  Masseters electrodes will be fixed parallel to the exocanthion-gonion line and with the upper pole of the electrode under the tragus-labial commissural line. Temporalis electrodes will be positioned along the anterior margin of the muscle (corresponding to the frontoparietal suture). Suprahyoid muscles electrodes will be placed in the submental area nearly 1 cm posterior to the mental symphysis, paramedian to the midline and lightly diverging. A reference electrode will be applied to the forehead of the patient.

SUMMARY:
Transverse maxillary constriction is a malocclusion that subsists when the distance between the upper first molars palatal cuspids is lower than the distance between the lower first molars vestibular center fossae. Consequently it can be clinically expressed with a narrow and high palatal vault, a unilateral or bilateral crossbite, dental crowding, and/or reduced volume of the nasal cavities.

It is one of the most common malocclusions in children, with a prevalence of 8 to 22% among orthodontic patients in primary and mixed dentition and 5 to 15% among the general population. The hypothesis of this study is that transverse maxillary constriction correction by Rapid Maxillary Expansor achieves improved muscles activation potential in treated patients and improved symmetry in patient with unilateral crossbite. The aim of this study is to evaluate electromyographic activity of the masseter, anterior temporalis and suprahyoid muscles in clentching, chewing and swallowing in patients undergoing expansion therapy of the maxillary with rapid palatal expander. The electromyographic evaluation is carried out before the treatment (T0), at the end of the expansion (T1) and after 6 months from T1 (T2).

DETAILED DESCRIPTION:
Transverse maxillary constriction subsists when the distance between upper first molars palatal cuspids is lower than the distance between lower first molars vestibular central fossae. It can be clinically expressed with a narrow and high palatal vault, a unilateral or bilateral crossbite, dental crowding and/or reduced volume of the nasal cavities. It is one of the most common malocclusions in children, with a prevalence of 8 to 22% among orthodontic patients in primary and mixed dentition and 5 to 15% among general population. The hypothesis of this study is that transverse maxillary constriction correction by Rapid Maxillary Expander (RME) affects masticatory muscles activation potential and improves activation symmetry in patient with unilateral crossbite. The aim of this study is to evaluate electromyographic activity of masseters, anterior temporalis and suprahyoid muscles in clenching, chewing and swallowing in patients undergoing maxillary expansion with RME. The electromyographic evaluation is carried out before treatment (T0), at the end of the expansion (T1) and 6 months later (T2). Detailed Description: Transverse maxillary constriction subsists when the distance between upper first molars palatal cuspids is lower than the distance between lower first molars vestibular central fossae. It can be clinically expressed with a narrow and high palatal vault, a unilateral or bilateral crossbite, dental crowding and/or reduced volume of the nasal cavities. It is one of the most common malocclusions in children, with a prevalence of 8 to 22% among orthodontic patients in primary and mixed dentition and 5 to 15% among general population. One of the most frequent expression of transverse maxillary constriction is unilateral crossbite, that consists in an inverted bucco-lingual relationship between one or more posterior teeth (canine to molars) with their antagonists; it can be present both in deciduous and permanent dentition. There is evidence that an altered relationship between upper and lower teeth is associated with asymmetric masticatory function that has been related to asymmetric contraction of masticatory muscles, decreased thickness of the cross-sided masseter muscle and altered masticatory pattern. This condition could lead to an asymmetric development of the mandibular bone during growth. Many authors conclude that early treatment of transverse maxillary constriction with RME would be recommended to reduce the risk of development of skeletal asymmetries and temporomandibular disorders (TMD). Muscle activity is commonly recorded by means of surface electromyography (sEMG). However sEMG data can be affected by various artifacts, resulting in questionable interpretation of the results. A standardisation procedure allows to reduce variability of the assessment of masticatory muscle activity during static and dynamic tasks.

- Page 2 of 6 [DRAFT] -

The hypotheses of this study are:

Patients with transverse maxillary constriction improve muscles activation potential after rapid maxillary expansion; correction of unilateral posterior crossbite by rapid maxillary expansion improves muscles activation potential symmetry.

The main objectives of this study are:

* to evaluate the activity of superficial masseters, anterior temporalis and suprahyoid muscles in patients with traverse maxillary constriction, using surface electromyography with a standardized protocol. The test consists of detecting muscles activity in maximum clenching (on cottons and on teeth), during swallowing and chewing;
* to evaluate whether the presence of unilateral posterior crossbite is associated with asymmetrical activation of superficial masseters, anterior temporalis and suprahyoid muscles;
* to compare intra-patient results before and after traverse maxillary constriction correction. The electromyograph that will be used is Easy-MYo EMG Tracer of 3 Technology Srl; Udine, Italy. It records muscular activity of superficial masseters, anterior temporalis and suprahyoid muscles. Disposable bipolar surface electrodes (21 × 41 mm, 20 mm inter-electrode distance; F3010; Fiab) will be used. The patient's skin will be clean with cotton gauze soaked in alcohol before electrodes placement to reduce skin impedance. The operator will palpate the muscle belly while the patient clenches his teeth and will position surface electrodes in parallel to muscular fibres.

Doing so the position of the electrodes results as follows:

Masseters electrodes will be fixed parallel to the exocanthion-gonion line and with the upper pole of the electrode under the tragus-labial commissural line. Temporalis electrodes will be positioned along the anterior margin of the muscle (corresponding to the frontoparietal suture). Suprahyoid muscles electrodes will be placed in the submental area nearly 1 cm posterior to the mental symphysis, paramedian to the midline and lightly diverging. A reference electrode will be applied on the forehead of the patient.

The sEMG analysis will be composed of four parts:

Masticatory muscle standardisation procedures (repeated thrice):

two 10mm thick cotton rolls will be positioned on the mandibular posterior teeth of each participant, and a 5 second maximum voluntary contraction will be recorded to standardize anterior temporalis and superficial masseters sEMG signals. The mean sEMG potential obtained in the first acquisition was set at 100%, and all further ssEMG potentials will be expressed as a percentage of this value (μV/μV × 100); Maximum voluntary teeth clenching: patients will be asked to clench their teeth in maximum intercuspation as hard as possible for 5 seconds.

Submental muscle standardisation procedures: participants will be asked to push their tongue against the palate (without teeth clenching), and a 5 seconds sEMG suprahyoid muscles activity will be recorded. All further sEMG potentials will be expressed as a percentage of this value (μV/μV × 100).

Saliva swallowing: participants will be asked to keep their mouth open to accumulate saliva and, when needed, to swallow "freely" (as usual) and a 5 seconds sEMG activity will be recorded.

Three EMG sessions will be recorded:

1. before starting treatment with Rapid Maxillary Expander (RME) (T0);
2. at the end of RME activation (T1), established by the clinician, generally looking for hypercorrection, that is contact between upper molar palatal cuspid and lower molar buccal cuspid.
3. after 6 months from T1 (T2).

ELIGIBILITY:
Inclusion Criteria:

* Transverse maxillary constriction
* Patients needing maxillary expansion with Rapid Maxillary Expander (RME)

Exclusion Criteria:

* Systemic diseases or congenital anomalies affecting craniofacial growth or development.
* Signs or symptoms of temporomandibular disorder (TMD).
* Dental pain.
* Previous orthopedic/orthodontic treatment/s.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Percentage Overlapping Coefficient - POC % | Baseline (T0), end of activations - approximately 14-30 days - (T1), after 6 months from T1 (T2)
  Indicates in % the ratio between the activation of the left muscle compared to the right one and its value is between 0 and 100%. A POC of 100% identifies two muscles that activate symmetrically. A lower value shows a greater asymmetry of muscles activation. There were 95% of subjects without muscular imbalances of dental origin who had POC values between 80 and 90% (Ferrario et al, 2000). The POC detected are: TA, MM and mean.
Change in Asymmetry index - ASIM % | Baseline (T0), end of activations - approximately 14-30 days - (T1), after 6 months from T1 (T2)
  It compares the influence of dental contacts on the total activity of the right MM and TA with respect to the left MM and TA. Its value varies between -100% and +100%. A negative value indicates a greater differential activity of the left muscles; conversely, a positive value indicates a greater differential activity of the right muscles. There was a total of 95% of subjects without muscular imbalances of dental origin having values of asymmetry between ± 10% (Ferrario et al, 2000);
Change in Activation Index - ATTIV % | Baseline (T0), end of activations- approximately 14-30 days - (T1), after 6 months from T1 (T2)
  It compares the influence of dental contacts on the TA activity in relation to MM activity. A negative value implies greater differential recruitment of TA, while a positive value implies greater differential recruitment of the MM. There was a total of 95% of subjects without muscular imbalances of dental origin having activation values between ± 10% (Ferrario et al, 2000);
Change in TORQUE % | Baseline (T0), end of activations- approximately 14-30 days - (T1), after 6 months from T1 (T2)
  Torque measures the differential activity of the right TA and left MM in relation to the antagonist torque. A prevalence of the right TA and left MM muscles, or right MM and left TA, may result in twisting forces on the jaw resulting in latero-deviation. This index ranges between -100% and +100%. -100% indicates the total prevalence of left TA and right MM, + 100% indicates the total prevalence of right TA and left MM. There was a total of 95% of subjects without muscular imbalances of dental origin having torque values between ±10% (Ferrario et al, 2000).
Change in IMPACT % | Baseline (T0), end of activations - approximately 14-30 days - (T1), after 6 months from T1 (T2)
  It quantifies the total muscular activity performed during MVC relative to the standardization clenching on cotton rolls.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Mac, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data are available upon motivated request to the Principal Investigator.